CLINICAL TRIAL: NCT01982708
Title: A Prospective Study of a Haptic Device Evaluation of the Acute Abdomen
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Robert Osmer, MSU Surgeon, Michigan State University
Other Study IDs: 13-744FM
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Acute Abdomen
Keywords: Evaluation
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesis is a haptic sensor can aid in the evaluation of the acute abdomen. Investigators from the MSU Department of Surgery in Collaboration with MSU Engineering are assessing the ability of a non invasive, optical device that is placed on a patients abdomen (much like an ultrasound transducer) to evaluate a patient with an acute abdominal presentation. Conditions such as appendicitis, cholecystitis, diverticulitis or small bowel obstruction will be examined with the haptic device. Data will be collected by the device and later compared to the abdominal findings recorded from an examination conducted by the principle investigator who is a surgeon. The surgeon will not have acess to data collected by the haptic sensor and therefore it will have no impact on the decision making process in the care of the patient. The impact on the individual patient will require obtaining a consent to participate in the study, a few minutes to place the device gently on the abdomen and collect the sensor data. There is no direct benefit to the patient by participating in the study. The potential for such a study may be to develop the technology to have a device that non-medical staff can use to collect patient data and transmit that data to a healthcare provider at another location.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the MSU Acute Care Surgery service for the evaluation of abdominal pain.

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department and inpatient referrals for general surgery evaluation for acute abdominal presentation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hardness of the abdominal wall | At intial presentation with abdominal pain

SECONDARY OUTCOMES:
temperature of the abdominal wall | At initial presentation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Osmer, M.D., Principal Investigator — MichiaganSU; Marc Basson, M.D., PhD, MBA, Study Chair — Michigan State University
Locations (1):
- Sparrow Hospital, Lansing, Michigan, United States